CLINICAL TRIAL: NCT04584593
Title: Pilot Study to Detect SARS-CoV-2 Virus in Sperm : a COVID-19 Study.
Brief Title: Pilot Study to Detect SARS-CoV-2 Virus in Sperm
Acronym: COVSPERM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/20/0202; 2020-A01610-39 (Other: ID-RCB)
Record Dates: First submitted 2020-10-12; First posted 2020-10-14 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: COVID19; SARS-CoV Infection; Semen
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SARV-Cov (Other): Men will give semen, saliva, urine and blood specimens
  Interventions: Biological: Sample

INTERVENTIONS:
Biological: Sample — Men will give semen, saliva, nasopharyngeal, urine and blood specimens

SUMMARY:
This is a prospective study involving 50 patients, with acute SARS-CoV-2 infection and a positive RNA detection. Men will give semen, saliva, urine and blood specimens following RT-PCR diagnosis and 15, 30, 60 and 90 days after. SARS-CoV-2 RNA will be detected in seminal plasma, native semen cells and processed spermatozoa.

The purpose of this study is to seek the presence of SARS-CoV-2 in semen, to determine its localization and infectiousness and to assess the efficiency of spermatozoa processing methods to obtain virus free spermatozoa.

DETAILED DESCRIPTION:
Since the end of 2019, an epidemic of SARS-CoV-2 infections (COVID-19) began in China and is now a global pandemic affecting more than 3 millions of people. Droplets and close contact are the most common routes of transmission of SARS-CoV-2 and aerosol transmission may be another route. Researchers have detected SARS-CoV-2 in samples of respiratory tract, saliva, stool, gastrointestinal tract, urine, tears and conjunctival secretions of COVID-19 patients.

Vertical transmission from mother to infant has been suspected, but not confirmed to date. Information about localization of SARS-CoV-2 in the genital tract or shedding is poorly documented and the results of these studies were discrepant. One of two studies have reported SARS-CoV-2 RNA in semen from six infected patients. However, there is no data on the duration of the seminal excretion of the virus, its viral load and infectiousness and on its localization in semen compartments (cells, seminal plasma, spermatozoa).

The purpose of this study is to seek the presence of SARS-CoV-2 in semen, to determine its localization and infectiousness and to assess the efficiency of spermatozoa processing methods to obtain virus free spermatozoa.

This is a prospective study involving 50 patients, with acute SARS-CoV-2 infection and a positive RNA detection. Men will give semen, saliva, urine and blood specimens following RT-PCR diagnosis and 15, 30, 60 and 90 days after. SARS-CoV-2 RNA will be detected in seminal plasma, native semen cells and processed spermatozoa.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 50, male.
* Patient in acute phase of infection with SARS-CoV-2 and whose RT-PCR shows the viral genome in the nasopharyngeal or salivary sample or in any other sample.
* Patient who can come to the laboratory for samples
* Patient having given his free and informed consent and having signed the consent
* Patient affiliated to a social security scheme or equivalent

Exclusion Criteria:

* Patient having previously consulted for male infertility or having previously carried out a semen examination which was abnormal (WHO standard)
* Patient with ejaculation disorder or unable to take a semen sample or with an abnormal semen volume (<1.5 mL).
* Patient who would present serious clinical signs that would not allow him to travel to the investigating center to take samples.
* Patient under a protection regime for adults (including guardianship, curatorship or safeguard of justice.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Semen sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 genomic RNA in patient sperm | 3 month
  Search for presence of SARS-CoV-2 genomic RNA in patients sperm when they are in the acute phase of the infection with reverse transcriptase polymerase chain reaction

SECONDARY OUTCOMES:
SARS-CoV-2 location in patient sperm | 3 month
  Search of location of SARS-Cov-2 in patient sperm after centrifugation

CONTACTS AND LOCATIONS:
Overall Officials: Louis BUJAN, PR, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Gallien S, Moro A, Lediguerher G, Catinot V, Paboeuf F, Bigault L, Berri M, Gauger PC, Pozzi N, Authie E, Rose N, Grasland B. Evidence of porcine epidemic diarrhea virus (PEDV) shedding in semen from infected specific pathogen-free boars. Vet Res. 2018 Jan 24;49(1):7. doi: 10.1186/s13567-018-0505-2. PMID 29368629
- [Background] Gallien S, Moro A, Lediguerher G, Catinot V, Paboeuf F, Bigault L, Gauger PC, Pozzi N, Berri M, Authie E, Rose N, Grasland B. Limited shedding of an S-InDel strain of porcine epidemic diarrhea virus (PEDV) in semen and questions regarding the infectivity of the detected virus. Vet Microbiol. 2019 Jan;228:20-25. doi: 10.1016/j.vetmic.2018.09.025. Epub 2018 Oct 11. PMID 30593368
- [Background] Baud D, Greub G, Favre G, Gengler C, Jaton K, Dubruc E, Pomar L. Second-Trimester Miscarriage in a Pregnant Woman With SARS-CoV-2 Infection. JAMA. 2020 Jun 2;323(21):2198-2200. doi: 10.1001/jama.2020.7233. PMID 32352491